CLINICAL TRIAL: NCT01619735
Title: Ureteroscopic Treatment of Intrarenal Stones - A Comparative Analysis of "Dusting" Versus "Basketing" With Holmium Laser Lithotripsy
Brief Title: "Dusting" Versus "Basketing" - Treatment Of Intrarenal Stones
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mitchell Humphreys, Consultant - Urology (surgical)/Associate Professor of Urology, Mayo Clinic
Other Study IDs: 12-002553
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Kidney Calculi; Kidney Stones; Nephrolithiasis; Renal Stones
Keywords: Kidney Calculi; Kidney Stones; Nephrolithiasis; Renal Stones
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fragments basketed: "Active" extraction is whereby the ureteroscope is passed back and forth into the kidney to remove all visible stone fragments.
- Fragments dusted: "Dusting" is whereby the stones are broken into tiny fragments or "dust" with the intention that achieving such a small stone size will allow the stones to pass spontaneously.

SUMMARY:
The purpose of this study is to evaluate outcomes of an established procedure for treatment of kidney stones that are present within the inner aspect of the kidney. This procedure is called flexible ureteroscopy, which involves placing a small camera through the urethra while anesthetized (asleep), up the ureter (the tube connecting kidney and bladder) and into the kidney to the kidney stone. Then, the stone is broken into tiny fragments using a small laser called a Holmium laser. While this treatment is a well-established option for treatment of these stones, there are several different techniques used to help eliminate them from the kidney. Some urologists treat the stone by a method called "active" extraction whereby the ureteroscope is passed back and forth into the kidney to remove all visible stone fragments. Others use a method called "dusting" whereby the stones are broken into tiny fragments or "dust" with the intention that achieving such a small stone size will allow the stones to pass spontaneously. There has not been a systematic and rigorous comparison of these techniques in terms of treatment outcomes. By collecting information on the success of treatment, the investigators hope to provide benchmark data for future studies of kidney stone treatment and improve the care of all patients who need surgery for their kidney stones.

The investigators hypothesize that the stone free rate for renal stone(s) 5-15 mm is around 90% and that the stone clearance rate with be 20% higher in those patients that undergo complete stone fragment extraction versus those that undergo stone dusting (residual fragments < 2mm).

DETAILED DESCRIPTION:
To date, there is inadequate literature to confidently determine the ideal technique of stone extraction during ureteroscopy, an endourologic procedure for the treatment of kidney stones. The goals of ureteroscopy for intrarenal stones are to fragment stones and minimize residual fragments while doing so in a safe and expeditious way with minimal harm to the patient. Options for the treatment of intrarenal stones consist of using a basket to pull them out or a laser to break them into small fragments. When stones are deemed too large to be basketed primarily, the standard preference in ureteroscopic laser lithotripsy is use of the Holmium:YAG laser which can effectively break stones into fragments small enough to remove or pass spontaneously.

There is no consensus on how to achieve optimal stone clearance once the primary stone is fragmented with lithotripsy. Many urologists choose to "dust" the stone by breaking it into tiny fragments < 1 - 2 mm in size with the assumption that stone fragments of such a small size will pass spontaneously after surgery. This can theoretically decrease operative times and lower risk of ureteral trauma by minimizing repetitive introduction and removal of the ureteroscope. Others choose to actively extract each possible stone fragment during the procedure thereby increasing the immediate stone-free outcome.

Active extraction however typically increases costs as it requires use of a basket or grasper and ureteral access sheath. To date, only one prospective, randomized study has addressed the practice of active extraction vs spontaneous passage, the results of which suggested higher rates of residual stone fragments, hospital readmissions and need for ancillary procedures when stones were not actively extracted (8). This study was criticized for not following a standardized operative protocol and not reporting several important outcomes including stone composition. Additionally, this study used semirigid ureteroscopy, specifically addressed ureteral rather than intrarenal stones, and did not follow a "dusting" protocol assuring minimal size of residual fragments.

Complete eradication of stone fragments is one of the primary outcomes of ureteroscopy as residual renal stone fragments after ureteroscopy have been shown to lead to a subsequent stone event in approximately 20% of cases(9). However, maximizing eradication of stone fragments must not come at the expense of the patient. For this reason it is important to consider the operative variables associated with the different techniques employed to clear stone during such procedures.

For example, an average of nearly three times as much laser energy was used to fragment the stone into tiny pieces compared to active extraction (8). Conversely, active extraction of stone fragments requires introducing and removing the ureteroscope through the ureter a greater number of times in order to facilitate stone removal; which generally requires use of a ureteral access sheath, a treatment with its own associated risk.(10). The short term and long term differences resulting from use of these techniques is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

* Radiopaque renal stones above the level of the ureteropelvic junction
* Kidney stones must range up to 20 mm in size or in the case of multiple stones the conglomerate diameter (additive maximal diameter of all stones on axial imaging of computed tomography) up to 20 mm is required for inclusion
* Patient must be a suitable operative candidate for flexible ureteroscopy

Exclusion Criteria:

* Patients who have had prior ipsilateral upper urinary tract reconstructive procedures or history of ipsilateral ureteral stricture
* Patients who have undergone prior radiotherapy to the abdomen or pelvis and those who have a neurogenic bladder or spinal cord injury
* Pregnant subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified at clinic visit or hospital admission
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2013-04; Primary Completion 2017-03-22 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
Stone-free rate | 4-6 weeks post-operatively
  To assess for stone-free rate using K.U.B. (kidney-ureter-bladder) plain radiograph and renal ultrasound. If there is a discrepancy in follow up imaging between the presence of residual stones or fragments between the KUB and renal ultrasound, the KUB will be considered the reference standard for small fragments less than 4mm unless the stone composition is uric acid. If fragments 5 mm or larger exist it will be up to the discretion of the surgeon to order a CT to better delineate the presence of residual stones and their impact on the clinical management of that patient.

SECONDARY OUTCOMES:
Stone recurrence rate | 12 months post operatively
  Stone recurrence rate one year after surgery
Retreatment rate | 12 months post operatively
  Evaluating the retreatment rate one year post operation

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Humphreys, MD, Principal Investigator — Mayo Clinic
Locations (9):
- United States (8):
  - Mayo Clinic, Scottsdale, Arizona
  - UCSD, San Diego, California
  - James Buchanan Brady Urological Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Bellevue Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University School of Medicine, Nashville, Tennessee
- University of British Columbia, Vancouver, British Columbia, Canada